CLINICAL TRIAL: NCT05255159
Title: Lesion-to-lesion Comparison of 68Ga-HA-DOTATATE, 18F-DOPA, and 18F-FDG PET/CT in the Evaluation of Metastatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREBA.CC-21-0353
Record Dates: First submitted 2022-01-31; First posted 2022-02-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DOPA PET/CT scan (Experimental): 4 MBq/kg (minimum 100 MBq, maximum 600 MBq) 18F-DOPA injected intravenously with 40 mg furosemide and subsequent whole body PET/CT scan
  Interventions: Diagnostic Test: 18F-DOPA with furosemide

INTERVENTIONS:
Diagnostic Test: 18F-DOPA with furosemide — Diagnostic 18F-DOPA PET/CT scan

SUMMARY:
This study is a single centre non-randomized non-blinded phase II prospective cohort study including 50 participants. The objective of this study is to directly compare 68Ga-HA-DOTATATE, 18F-DOPA, and 18F-FDG activity in patients with metastatic neuroendocrine tumors (NETs) on a lesion-by-lesion basis. The investigators will determine the prevalence of concordant versus discordant disease. Secondary objectives include assessing the standardized uptake value (SUV) and determining if there is any correlation between discordance and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy proven neuroendocrine tumor including (but not limited to): gastrointestinal NET, pancreatic NET, pulmonary NET, NET unknown primary, pheochromocytoma, paraganglioma, medullary thyroid cancer, medulloblastoma, meningioma
* At least two abnormal 68Ga-HA-DOTATATE positive lesions suspected to represent neuroendocrine tumor (at least tow lesions with SUVmax > SUV meanliver).
* Age greater or equal to 40
* Ability to provide written informed consent prior to participation in the study

Exclusion Criteria:

* Weight > 225 kg (weight limitation of PET/CT scanner)
* Inability to scan (ie. extreme claustrophobia) or inability to lie still for imaging
* Any medical condition, serious inter-current illness, or other extenuating circumstance that, in the opinion of the investigator or attending department physician, may significantly interfere with study performance or interpretation
* Previous allergic reaction to 18F-DOPA
* Lack of intravenous access
* Pregnant
* Breastfeeding
* Less than 40 years old

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Lesion-to-lesion comparison of activity on 68Ga-HA-DOTATATE, 18F-DOPA, and 18F-FDG PET/CT scans | Within 1 year after completion of both 18F-DOPA and 18F-FDG PET/CT scans
  Participants will be categorized as having concordant disease (all lesions 68Ga-HA-DOTATATE avid) or discordant disease (one or more lesions not 68Ga-HA-DOTATATE avid).

SECONDARY OUTCOMES:
SUV of lesions on 68Ga-HA-DOTATATE, 18F-DOPA, and 18F-FDG PET/CT scans | Within 1 year after completion of both 18F-DOPA and 18F-FDG PET/CT scans
  SUVmax of all lesions on all scans will be recorded and compared to SUVmean of the liver and blood pool
Assessment of disease progression - 12 months | 12 months after completion of the 68Ga-HA-DOTATATE, 18F-FDG, and investigational 18F-DOPA PET/CT scans
  All available clinical information will be reviewed 12 months after completion of the PET/CT scans with expert determination of treatment response, no treatment response, or disease progression
Assessment of disease progression - 18 months | 18 months after completion of the 68Ga-HA-DOTATATE, 18F-FDG, and investigational 18F-DOPA PET/CT scans
  All available clinical information will be reviewed at 18 months after completion of the PET/CT scans with expert determination of treatment response, no treatment response, or disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Abele, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No